CLINICAL TRIAL: NCT04352647
Title: Observational Study on the Prevalence of Urinary Incontinence in Federates Athletes in Castilla y León.
Brief Title: Observational Study on the Prevalence of Urinary Incontinence in Federates Athletes.
Status: Completed | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Other Study IDs: 003/2020
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Urinary Incontinence
Keywords: Women health; Sports; Incontinence, urinary stress
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- female athletes over the age of 18: the presence or absence of urinary incontinence in female athletes is studied. In addition, the quality of life and other aspects are evaluated
  Interventions: Behavioral: female athletes

INTERVENTIONS:
Behavioral: female athletes — The type of incontinence is assessed, whether there are risk factors and quality of life and psychological performance

SUMMARY:
To study the prevalence of urinary incontinence (UI) in female athletes from Castilla y León, as well as the category of athletics with the highest number of losses, the most incident risk factors and the bio-psycho-social consequences that it leads to.

DETAILED DESCRIPTION:
Elaboration of a survey, based on two validated questionnaires to which 63 participants have answered, to carry out an analytical, transversal and observational study. All the participants are women, of age, federated in athletics and belonging to Castilla y León.

UI has a high prevalence (44.4%) in female athletes, being more common in those who practice long-distance races. As age and years of sport increase, the incidence of this pathology increases. Absorbent pads are used by more than half of the incontinent women, while the rest wet their underwear. Menopause, childbirth and surgery in the region are risk factors for UTIs, while the presence of urinary tract infections or candidiasis are not. The results affirm that urine leaks do not cause anxiety or depression, but they do affect your sporting life.

ELIGIBILITY:
Inclusion Criteria:

* Female sex.
* Adulthood.
* Federated in athletics.

Exclusion Criteria:

* Men.
* Those women who are no longer federated or who are minors.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: female athletes over 18 and under 65
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants suffering from urinary incontinence | 2 months
  observe whether female athletes suffer from urinary incontinence

SECONDARY OUTCOMES:
Number of participants suffering from urinary incontinence with a bio-psycho-social component | 2 months
  observe the bio-psycho-social component of suffering from urinary incontinence
Incidence rate and urinary incontinence according to athletic discipline | 2 months
  to see if athletic discipline is related to urinary incontinence
Incidence rate and urinary incontinence and associated risk factors | 2 months
  look at the risk factors associated with urinary incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bo K, Berghmans LC. Nonpharmacologic treatments for overactive bladder-pelvic floor exercises. Urology. 2000 May;55(5A Suppl):7-11; discussion 14-6. PMID 10767443
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] MacLennan AH, Taylor AW, Wilson DH, Wilson D. The prevalence of pelvic floor disorders and their relationship to gender, age, parity and mode of delivery. BJOG. 2000 Dec;107(12):1460-70. doi: 10.1111/j.1471-0528.2000.tb11669.x. PMID 11192101
- [Background] Turner CE, Young JM, Solomon MJ, Ludlow J, Benness C. Incidence and etiology of pelvic floor dysfunction and mode of delivery: an overview. Dis Colon Rectum. 2009 Jun;52(6):1186-95. doi: 10.1007/DCR.0b013e31819f283f. PMID 19581867
- [Background] Wohlrab KJ, Rardin CR. Impact of route of delivery on continence and sexual function. Clin Perinatol. 2008 Sep;35(3):583-90, xii. doi: 10.1016/j.clp.2008.06.001. PMID 18952024
- [Background] Haakstad LAH, Gjestvang C, Lamerton T, Bo K. Urinary incontinence in a fitness club setting-is it a workout problem? Int Urogynecol J. 2020 Sep;31(9):1795-1802. doi: 10.1007/s00192-020-04253-0. Epub 2020 Mar 4. PMID 32130465
- [Background] Hay-Smith J, Morkved S, Fairbrother KA, Herbison GP. Pelvic floor muscle training for prevention and treatment of urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD007471. doi: 10.1002/14651858.CD007471. PMID 18843750
- [Background] Titman SC, Radley SC, Gray TG. Self-management in women with stress incontinence: strategies, outcomes and integration into clinical care. Res Rep Urol. 2019 Apr 17;11:111-121. doi: 10.2147/RRU.S177826. eCollection 2019. PMID 31114767
- [Derived] Velazquez-Saornil J, Mendez-Sanchez E, Gomez-Sanchez S, Sanchez-Mila Z, Cortes-Llorente E, Martin-Jimenez A, Sanchez-Jimenez E, Campon-Chekroun A. Observational Study on the Prevalence of Urinary Incontinence in Female Athletes. Int J Environ Res Public Health. 2021 May 24;18(11):5591. doi: 10.3390/ijerph18115591. PMID 34073782
- See also: incontinence urinary — http://scielo.isciii.es/scielo.php?script=sci_abstract&pid=S1137-66272006000300006
- See also: incontinence urinary — http://www.medicapanamericana.com/libro/campbell-walsh-urologia-wein-10-edicion-tomo-2